CLINICAL TRIAL: NCT06784297
Title: INTERMEDIATE-SIZE PATIENT POPULATIONS EXPANDED ACCESS to TREATMENT for SARCOPENIC OBESITY
Acronym: STEM-META-EAP
Status: Temporarily not available | Type: Expanded Access
Sponsor: Immunis, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: STEM-META-EAP
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-01-21 (Actual); Status verified 2025-01

CONDITIONS: Sarcopenia; Obesity and Obesity-related Medical Conditions
MeSH Terms: conditions — Sarcopenia; Obesity

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Biological: IMM01-STEM — The individuals receiving expanded access will receive a treatment identical to the most convenient regimen in the current clinical trial (STEM-META). The treatment will consist of one i.m. injection per week containing 2 mg of total protein in 2 mL, for a total of 4 weeks (4 injections). As more efficacy information accumulates, the treatment plan will be adjusted accordingly to maximize the potential benefit.

SUMMARY:
The expanded access is designed for patients requesting the treatment, and whose medical condition may benefit from treatment, but are unable to participate in any other IMM01-STEM clinical trial in their physician's opinion for reasons that include: (1) They do not meet enrollment criteria, or (2) They cannot perform the assessment of outcomes, or (3) The trial site is not geographically accessible.

ELIGIBILITY:
Inclusion Criteria:

1. Sex: male or post-menopausal female (as defined by the absence of a period for at least 12 consecutive months)
2. Race/nationality: all races and ethnicities accepted for which there are validated reference values for obesity and sarcopenia diagnostic criteria
3. Disease characteristics: to be eligible, the participant must meet one criterion for obesity and at least one criterion for sarcopenia, as defined below:

Obesity:

1. Abdominal obesity defined by a waist circumference ≥ 40 inches (102 cm) for men, ≥ 35 inches (88 cm) for women (American Heart Association)
2. Abdominal obesity as a waist-to-hip ratio of at least 0.90 in men and 0.85 or more for
3. No obesity, normal BMI women (World Health Organization)

Sarcopenia:

i) Grip strength: < 16 kg (women), < 27 kg (men) in the dominant hand, or, ii) Gait speed < 0.8 m/s (men and women) iii) Clinical evidence of sarcopenia alternative to grips strength and gait speed measurements, as judged by the physician

Exclusion Criteria:

1. Qualifying individuals by the current enrollment criteria that are in a 50-mile geographical radius of any IMM01-STEM clinical trial site or a potential clinical site.
2. Inability to sign an informed consent
3. Concomitant investigational drugs and treatments
4. Concomitant medication included in the table 1.
5. Current malignancy or recent malignancy in complete remission less than 3 years
6. BMI < 20
7. Major surgical procedures in the past 30 days.
8. Cognitive impairment, Alzheimer disease,
9. Progressive autoimmune disorders including rheumatoid arthritis, muscular dystrophy, multiple sclerosis, systemic sclerosis, inclusion body myositis, idiopathic inflammatory myopathy, and similar conditions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult